CLINICAL TRIAL: NCT04577417
Title: Stimulant Medication Effects on Auditory Sensitivity and Acoustic Reflex in Adolescents With ADHD
Brief Title: Stimulant Medication Effects on Auditory Sensitivity in Teens With ADHD
Status: Completed | Type: Observational
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 1600804
Record Dates: First submitted 2020-09-18; First posted 2020-10-06 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Attention Deficit Hyperactivity Disorder; Attention Deficit Disorder; Attention Deficit Disorder With Hyperactivity
Keywords: stimulant medication
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Amphetamine; Dexmethylphenidate Hydrochloride; Dextroamphetamine; Methylphenidate; Adderall; Lisdexamfetamine Dimesylate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- ADHD: Adolescents, male or female, ages 13-19, diagnosed with ADHD, all subtypes, based on the fifth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) and under treatment with a stimulant medication with the same drug and dosage for at least 12 months before their study participation date
  Interventions: Drug: ADHD stimulants, for example, amphetamine, dexmethylphenidate, dextroamphetamine, methylphenidate
- Control: Adolescents, male or female, ages 13-19, with normal health status and development

INTERVENTIONS:
Drug: ADHD stimulants, for example, amphetamine, dexmethylphenidate, dextroamphetamine, methylphenidate — Both ADHD and control groups of subjects will participate in 2 sessions (on-med and off-med conditions) conducted on the same day. ADHD group will be asked to come to the laboratory in the morning before taking their morning ADHD stimulant medication. They will be tested before and after taking their ADHD medication (off-med and on-med conditions). The investigators will observe changes between the two conditions.
  Other Names: Adderall; Focalin; Ritalin; Vyvanse; Concerta
  Groups: ADHD

SUMMARY:
The aims of this study are to evaluate auditory sensitivity in teenagers with ADHD using acoustic reflex thresholds (ART) and to examine the effects of ADHD stimulant medication on ART.

DETAILED DESCRIPTION:
Attention-deficit/hyperactivity disorder (ADHD) is the most common neurodevelopmental disorder in children. Besides core ADHD symptoms (inattentiveness, hyperactivity, impulsivity), ADHD also affects the ability to perceive and process sounds. Both hypersensitivity and hyposensitivity to loud sounds are common symptoms in ADHD patients. With stimulant medication, individuals with ADHD become more tolerant of loud noise than when they were non-medicated. It remains unknown exactly how stimulant medication alters the loudness perception. The proposed study will use the acoustic reflex to objectively measure auditory sensitivity to loud sounds. The aims of this study are to evaluate auditory sensitivity in patients with ADHD using acoustic reflex thresholds (ART) and to examine the effects of ADHD stimulant medication on ART. Eligible participants will participate in two sessions (off-med and on-med conditions) conducted on the same day. ADHD patients will be asked to come to the laboratory before taking their ADHD medication. The investigators will repeat three tests before and after taking stimulant medication. The investigators will also conduct screening tests during and between the first and second sessions. The investigators will compare a difference between the two independent groups (ADHD vs. Control) and compare a within subject difference between medication conditions (on-med vs. off-med).

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for all:

* Participant must be aged 13 to 19 years
* Males and females
* All ethnicities
* All socioeconomic statuses
* Normal hearing
* English as a primary language

Additional inclusion criteria for ADHD group:

* Participants must meet diagnostic criteria for attention-deficit/hyperactivity disorder (ADHD), all subtypes, based on the fifth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5)
* Stimulant medication with the same drug and dosage for at least 1 year before their enrollment date

Exclusion Criteria:

* History of any major neurological disorders (e.g. seizures excluding febrile seizure under age 6 years, tumors, brain injury, cerebral palsy, tic disorders)
* History of any other major neuropsychiatric disorders (e.g. autism spectrum disorder, mood dysregulation),
* Presence of pressure equalization tubes in either ear
* Documented hearing impairment 20 decibel or higher hearing loss in either ear
* Estimated low cognitive function based on the NIH Toolbox Cognition age-corrected scores (<70)

Additional exclusion criteria for the ADHD group

* Treatment with any psychotropic medications other than stimulants
* Treatment with any ADHD medication other than stimulants (e.g. alpha-agonists, norepinephrine reuptake inhibitors)

Additional exclusion criteria for the control group

• Treatment with any psychotropic medication

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescents with ADHD and typically developing adolescents
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2020-09-13 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Acoustic reflex | through study completion, an average of 1 year
  Acoustic reflex thresholds in each ear
Loudness discomfort level | through study completion, an average of 1 year
  Average loudness levels judged as uncomfortably loud sounds by each participant
Speech perception in noise | through study completion, an average of 1 year
  Speech perception scores in each ear measured in two separate sessions

SECONDARY OUTCOMES:
Tympanogram | through study completion, an average of 1 year
  Results of tympanometry (type, volume, pressure, compliance, gradient) to measure middle ear function
Otoacoustic emissions | through study completion, an average of 1 year
  Measure of inner ear function
NIH Toolbox Cognition testing | through study completion, an average of 1 year
  Measures of cognitive functions
Hearing screening | through study completion, an average of 1 year
  Pure-tone hearing test to measure hearing sensitivity
Sensory profile questionnaire | through study completion, an average of 1 year
  Sensory processing assessment
Fidgeting | through study completion, an average of 1 year
  Measure of wrist movements during the testing

CONTACTS AND LOCATIONS:
Overall Officials: Kyoko Nagao, PhD, Principal Investigator — Nemours
Locations (1):
- Nemours Children's Health, Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sydenstricker S, Moore A, Nagao K. Comparison of Fidgeting in Adolescents with Attention-Deficit/Hyperactivity Disorder Between Before and After Stimulant Medication Intake. J Child Adolesc Psychopharmacol. 2023 May;33(4):143-148. doi: 10.1089/cap.2022.0080. Epub 2023 Mar 10. PMID 36913518
- See also: Teenagers with ADHD may perceive loud sounds in a different way. Acoustical Society of America Press Room. — https://acoustics.org/2ppp8-teenagers-with-adhd-may-perceive-loud-sounds-in-a-different-way-alexandra-moore/